CLINICAL TRIAL: NCT01201837
Title: CHI SQUARE: Can HDL Infusions Significantly Quicken Atherosclerosis Regression? A Phase II, Multi-Center, Double-Blind, Ascending Dose, Placebo-Controlled, Dose-Finding Trial of CER-001 or Placebo in Subjects With Acute Coronary Syndrome
Brief Title: Effect of CER-001 on Atherosclerosis in Acute Coronary Syndrome (ACS) Patients - Efficacy and Safety: The CHI SQUARE Trial
Acronym: CHI SQUARE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cerenis Therapeutics, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CER-001-CLIN-002
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; HDL mimetic; ApoA-I
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — CER-001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Low Dose (Experimental): CER-001 Low Dose
  Interventions: Drug: CER-001
- Mid Dose (Experimental): CER-001 Mid Dose
  Interventions: Drug: CER-001
- High Dose (Experimental): CER-001 High Dose
  Interventions: Drug: CER-001

INTERVENTIONS:
Drug: Placebo — Weekly injection
  Arms: Placebo
Drug: CER-001 — Weekly injection
  Arms: High Dose; Low Dose; Mid Dose

SUMMARY:
Cardiovascular disease remains the most pressing healthcare issue for developed countries and is becoming so for developing countries. There are a number of chronic therapies available for long-term management of risk. Short term therapies for subjects with an acute event, such as an episode of acute coronary syndrome (ACS), are focused on reperfusion and removing thrombus but most subsequent events are caused by atherosclerotic plaque rupture at a different site. There are no approved therapies that can rapidly reduce the burden of unstable, inflamed plaque in the overall coronary vascular bed. HDL has multiple actions that could lead to atherosclerotic plaque stabilization, such as rapid removal of large quantities of cholesterol from the vasculature, improvement in endothelial function, protection against oxidative damage and reduction in inflammation. This study will assess the effects of CER-001, an ApoA-I-based HDL mimetic, on indices of atherosclerotic plaque progression and regression as assessed by intravascular ultrasound (IVUS) measurements in patients with (ACS).

ELIGIBILITY:
Inclusion Criteria:

* Male or female less than 75 years of age
* Acute coronary syndrome (acute chest pain and a diagnosis of ST segment elevation myocardial infarction, non-ST elevation myocardial infarction or unstable angina)
* Angiographic evidence of coronary artery disease with suitable "target" coronary artery for IVUS evaluation

Exclusion Criteria:

* Females of child-bearing potential
* Weight >120 kg
* Angiographic evidence of >50% stenosis of the left main artery
* Uncontrolled diabetes (HbA1C>10%)
* Hypertriglyceridemia (>500 mg/dL)
* Congestive heart failure (NYHA class III or IV)
* Ejection fraction <35%
* Uncontrolled hypertension (SBP >180 mm Hg)
* Known major hematologic, renal, hepatic, metabolic, gastrointestinal or endocrine dysfunction

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in Total Plaque Volume | Baseline and 3 weeks post final dose
  Absolute change in total plaque volume, as assessed by IVUS, from the baseline measurement to the follow-up taken ~3 weeks following the final dose of study medication (approximately 9 weeks after the baseline assessment)

SECONDARY OUTCOMES:
Percent Change in Plaque Volume | Baseline and 3 weeks post final dose
  Percent change in total plaque volume, as assessed by IVUS, from the baseline measurement to the follow-up taken ~3 weeks following the final dose of study medication (approximately 9 weeks after the baseline assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, MD, Principal Investigator — Montreal Heart Institute
Locations (47):
- United States (24):
  - Heart Center Research LLC, Huntsville, Alabama
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - VA San Diego Health Care Center, San Diego, California
  - Palm Beach Heart Institute, LLC - Zasa Clinical Research, Boynton Beach, Florida
  - Heart and Vascular Institute of Florida, Clearwater, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Saint Joseph Research Institute, Atlanta, Georgia
  - The Care Group, LLC, Indianapolis, Indiana
  - Suburban Hospital, Bethesda, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Detroit Medical Center (DMC) Cardiovascular Institute, Detroit, Michigan
  - Cardiac and Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Alegent Research Center, Omaha, Nebraska
  - Buffalo Heart Group, Buffalo, New York
  - Buffalo Cardiology & Pulmonary Associates, Williamsville, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Sanford Heart Center, Fargo, North Dakota
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Sanford Research / USD, Sioux Falls, South Dakota
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Dallas VA Medical Center, Dallas, Texas
  - MultiCare Health System Research Institute / Cardiac Study Center, Tacoma, Washington
- Canada (11):
  - Foothills Medical Centre, Calgary, Alberta
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - St. John Health Center, St. John's, Newfoundland and Labrador
  - London Health Sciences Center, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Centre de Santé et de Services Sociaux de Laval, Laval, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Montreal General Hospital Research Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie et Pneumologie de Québec (IUCPQ), Québec, Quebec
  - CSSS du Nord de Lanaudière, Saint-Charles-Borromée, Quebec
  - Centre Hospitalier Régional de Trois-Rivières, Trois-Rivières, Quebec
- France (3):
  - Hôpital Cardiologique du Haut-Lévesque, Bordeaux, Pessac Cedex
  - Clinique Pasteur, Toulouse
  - Centre Hospitalier Universitaire de Toulouse Rangueil, Toulouse
- Netherlands (9):
  - Onze Lieve Vrouwe Gasthius, Amsterdam, AC
  - Medisch Centrum Leeuwarden, Leeuwarden, AD
  - Medisch Centrum Alkmaar, Alkmaar, Amsterdam
  - Academic Medical Center, Amsterdam, AZ
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein, CM
  - Maassstadziekenhuis Cardiology Research, Rotterdam, DZ
  - Catharina Ziekenhuis Eindhoven, Eindhoven, EJ
  - Medisch Spectrum Twente, Enschede, ER
  - Canisius Wilhelmina Ziekenhuis, Nijmegen, SZ

REFERENCES:
- [Background] Nanjee MN, Doran JE, Lerch PG, Miller NE. Acute effects of intravenous infusion of ApoA1/phosphatidylcholine discs on plasma lipoproteins in humans. Arterioscler Thromb Vasc Biol. 1999 Apr;19(4):979-89. doi: 10.1161/01.atv.19.4.979. PMID 10195926
- [Background] Eriksson M, Carlson LA, Miettinen TA, Angelin B. Stimulation of fecal steroid excretion after infusion of recombinant proapolipoprotein A-I. Potential reverse cholesterol transport in humans. Circulation. 1999 Aug 10;100(6):594-8. doi: 10.1161/01.cir.100.6.594. PMID 10441095
- [Background] Spieker LE, Sudano I, Hurlimann D, Lerch PG, Lang MG, Binggeli C, Corti R, Ruschitzka F, Luscher TF, Noll G. High-density lipoprotein restores endothelial function in hypercholesterolemic men. Circulation. 2002 Mar 26;105(12):1399-402. doi: 10.1161/01.cir.0000013424.28206.8f. PMID 11914243
- [Background] Nieuwdorp M, Vergeer M, Bisoendial RJ, op 't Roodt J, Levels H, Birjmohun RS, Kuivenhoven JA, Basser R, Rabelink TJ, Kastelein JJ, Stroes ES. Reconstituted HDL infusion restores endothelial function in patients with type 2 diabetes mellitus. Diabetologia. 2008 Jun;51(6):1081-4. doi: 10.1007/s00125-008-0975-2. Epub 2008 Apr 4. No abstract available. PMID 18389214
- [Background] Drew BG, Duffy SJ, Formosa MF, Natoli AK, Henstridge DC, Penfold SA, Thomas WG, Mukhamedova N, de Courten B, Forbes JM, Yap FY, Kaye DM, van Hall G, Febbraio MA, Kemp BE, Sviridov D, Steinberg GR, Kingwell BA. High-density lipoprotein modulates glucose metabolism in patients with type 2 diabetes mellitus. Circulation. 2009 Apr 21;119(15):2103-11. doi: 10.1161/CIRCULATIONAHA.108.843219. Epub 2009 Apr 6. PMID 19349317
- [Background] Shaw JA, Bobik A, Murphy A, Kanellakis P, Blombery P, Mukhamedova N, Woollard K, Lyon S, Sviridov D, Dart AM. Infusion of reconstituted high-density lipoprotein leads to acute changes in human atherosclerotic plaque. Circ Res. 2008 Nov 7;103(10):1084-91. doi: 10.1161/CIRCRESAHA.108.182063. Epub 2008 Oct 2. PMID 18832751
- [Background] Waksman R, Torguson R, Kent KM, Pichard AD, Suddath WO, Satler LF, Martin BD, Perlman TJ, Maltais JA, Weissman NJ, Fitzgerald PJ, Brewer HB Jr. A first-in-man, randomized, placebo-controlled study to evaluate the safety and feasibility of autologous delipidated high-density lipoprotein plasma infusions in patients with acute coronary syndrome. J Am Coll Cardiol. 2010 Jun 15;55(24):2727-35. doi: 10.1016/j.jacc.2009.12.067. PMID 20538165
- [Background] Tardif JC, Gregoire J, L'Allier PL, Ibrahim R, Lesperance J, Heinonen TM, Kouz S, Berry C, Basser R, Lavoie MA, Guertin MC, Rodes-Cabau J; Effect of rHDL on Atherosclerosis-Safety and Efficacy (ERASE) Investigators. Effects of reconstituted high-density lipoprotein infusions on coronary atherosclerosis: a randomized controlled trial. JAMA. 2007 Apr 18;297(15):1675-82. doi: 10.1001/jama.297.15.jpc70004. Epub 2007 Mar 26. PMID 17387133
- [Background] Nissen SE, Tsunoda T, Tuzcu EM, Schoenhagen P, Cooper CJ, Yasin M, Eaton GM, Lauer MA, Sheldon WS, Grines CL, Halpern S, Crowe T, Blankenship JC, Kerensky R. Effect of recombinant ApoA-I Milano on coronary atherosclerosis in patients with acute coronary syndromes: a randomized controlled trial. JAMA. 2003 Nov 5;290(17):2292-300. doi: 10.1001/jama.290.17.2292. PMID 14600188
- [Derived] Tardif JC, Ballantyne CM, Barter P, Dasseux JL, Fayad ZA, Guertin MC, Kastelein JJ, Keyserling C, Klepp H, Koenig W, L'Allier PL, Lesperance J, Luscher TF, Paolini JF, Tawakol A, Waters DD; Can HDL Infusions Significantly QUicken Atherosclerosis REgression (CHI-SQUARE) Investigators. Effects of the high-density lipoprotein mimetic agent CER-001 on coronary atherosclerosis in patients with acute coronary syndromes: a randomized trial. Eur Heart J. 2014 Dec 7;35(46):3277-86. doi: 10.1093/eurheartj/ehu171. Epub 2014 Apr 29. PMID 24780501